CLINICAL TRIAL: NCT06360965
Title: A Randomized Controlled Trial on the Clinical Efficacy and Safety of Warm Meridians and Relieve Pain Plaster in Improving the Sequelae of Pelvic Inflammatory Disease and Chronic Pelvic Pain (Cold Dampness Stasis Type).
Brief Title: Clinical Trial of Acupoint Application in Improving the Sequelae of Pelvic Inflammatory Disease and Chronic Pelvic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Shoufa2024-3-7045
Record Dates: First submitted 2024-04-01; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Pelvic Inflammatory Disease; Chronic Pelvic Pain Syndrome
Keywords: Pelvic Inflammatory Disease; Chronic Pelvic Pain Syndrome; acupoint application; cold dampness stasis type
MeSH Terms: conditions — Pelvic Inflammatory Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Improved warm meridians and relieve pain plaster group (Active Comparator): Use an improved warm meridians and relieve pain plaster (about 7cm wide, 10cm long, and 0.5mm thick) to apply to the navel.
  Interventions: Drug: Improved warm meridians and relieve pain plaster
- Traditional warm meridians and relieve pain plaster group (Active Comparator): Select Angelica sinensis, Ligusticum chuanxiong, Cinnamon, Sichuan pepper, Corydalis yanhusuo, Fructus Evodiae, Paeonia lactiflorus, Artemisia argyi, Cyperus, Zelan, and Muxiang, mix in a ratio of 1.5:1:1.8:1.5:1.2:0.5:1.5:0.8:1.5:1.5, and use a grinder to grind and sieve; Take an appropriate amount of Vaseline and mix thoroughly with the above-mentioned powder in a 1:1 ratio. Take an appropriate amount of medication and place it in the center of the acupoint patch (8cm x 8cm). Press the medication evenly into a circular hole with a diameter of about 4cm and a depth of about 3mm, and align the patch.
  Interventions: Drug: Traditional warm meridians and relieve pain plaster
- Placebo plaster group (Placebo Comparator): Take an appropriate amount of Vaseline and mix thoroughly with 1% of the original ingredient, starch, and pigment. Take an appropriate amount of medication and place it in the center of the acupoint patch (8cm x 8cm). Press the medication evenly into a circular hole with a diameter of about 4cm and a depth of about 3mm, and align the patch.
  Interventions: Drug: Placebo plaster

INTERVENTIONS:
Drug: Improved warm meridians and relieve pain plaster — Starting from the 1st to 3rd day after the menstrual cycle is clean, apply it 6-8 hours before bedtime every day, with one day off. Apply 10 times per menstrual cycle as one course of treatment, with two consecutive courses of treatment.
  Arms: Improved warm meridians and relieve pain plaster group
Drug: Traditional warm meridians and relieve pain plaster — The treatment course is the same as the improved warm meridians and relieve pain plaster group.
  Arms: Traditional warm meridians and relieve pain plaster group
Drug: Placebo plaster — The treatment course is the same as the improved warm meridians and relieve pain plaster group.
  Arms: Placebo plaster group

SUMMARY:
Chronic Pelvic Pain is one of the common gynecological symptoms, characterized by persistent and non periodic pain in the pelvic cavity and surrounding tissues. It is often seen as a sequelae of pelvic inflammatory diseases caused by the failure to receive timely and correct treatment. This study compares the effectiveness of warm meridians and relieve pain plaster in relieving the sequelae of pelvic inflammatory disease and chronic pelvic pain symptoms, and evaluates the safety of improved patches and traditional patches, further promoting it to community grassroots hospitals.

DETAILED DESCRIPTION:
Chronic Pelvic Pain is one of the common gynecological symptoms, characterized by persistent and non periodic pain in the pelvic cavity and surrounding tissues. It is often seen as a sequelae of pelvic inflammatory diseases caused by the failure to receive timely and correct treatment. Chronic pelvic pain is mainly characterized by lower abdominal or lumbosacral pain, which may be accompanied by increased vaginal discharge. This disease has the characteristics of high incidence rate, long course, lingering, difficult to heal, easy to relapse, etc., which seriously affects women's reproductive health and quality of life, and increases the family and socio-economic burden. At present, there is no effective treatment method in Western medicine for the sequelae of pelvic inflammatory diseases and chronic pelvic pain, mainly targeting the symptoms of patients for treatment. Therefore, this study selected 102 patients with pelvic inflammatory disease sequelae and chronic pelvic pain (cold dampness stasis type) who met the inclusion criteria as the research subjects. They were randomly divided into an improved warm meridians and relieve pain plaster group, a traditional warm meridians and relieve pain plaster group, and a placebo group. Three groups of acupoint patches were applied to the navel, and the therapeutic effect was evaluated after two consecutive menstrual cycles. Follow up was conducted at the end of one menstrual cycle after the treatment, and adverse events during the research process were recorded. Compare the effectiveness of warm meridians and relieve pain plaster in relieving symptoms of this disease, and evaluate the safety of improved patches and traditional patches, further promoting it to community grassroots hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria of traditional Chinese and Western medicine for sequelae of pelvic inflammatory disease and chronic pelvic pain;
2. Transvaginal ultrasound examination shows thickening of the fallopian tube wall and fluid accumulation in the lumen, which may be accompanied by pelvic free fluid or fallopian tube ovarian masses;
3. The age range is 18-50 years old, married or with a history of sexual activity;
4. Those with a menstrual cycle of 21-35 days;
5. 4 points ≤ Pain Visual Analog Scale (VAS) < 7 points;
6. Those who have signed an informed consent form and are willing to receive treatment.

Exclusion Criteria:

1. Female patients who have fertility requirements during pregnancy, lactation, or in the short term;
2. Patients with gynecological diseases such as organic lesions of the reproductive system or gynecological acute abdomen;
3. Chronic pelvic pain caused by gynecological tumors, endometriosis, pelvic congestion syndrome, uterine fibroids, tuberculous pelvic inflammatory disease, and other diseases confirmed through examination;
4. Those with severe diseases such as cardiovascular, cerebrovascular, liver and kidney function, and digestive system;
5. Individuals with mental abnormalities and psychological disorders;
6. Individuals with allergic constitution or known allergies to the drugs and their components used in this experiment;
7. Patients currently participating in clinical trials of other drugs;
8. Other methods of treatment have already been or are currently being carried out, which may affect the indicators observed in this study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Main symptoms (lower abdominal pain) improvement level (visual analogue scale) | The baseline period, the treatment two menstrual cycle (about 8 weeks) and the follow-up period (about 12 weeks).
  Using the Visual Analog Scale (VAS), draw a 10cm thick straight line on the patient record card, with one end indicating no pain and the other end indicating unbearable severe pain. Patients should mark a point on the line based on the degree of lower abdominal pain (bloating or stabbing) they experience. Researchers use a straightedge to measure the straight-line distance from the starting point to the patient's designated point, and express the intensity of pain using the measured numbers. Record the specific mm measured by the patient.

SECONDARY OUTCOMES:
TCM syndrome score scale | The baseline period, the treatment two menstrual cycle (about 8 weeks) and the follow-up period (about 12 weeks) .
  The TCM syndrome score scale consists of three main symptoms and nine secondary symptoms. The main symptoms included abdominal pain, lumbosacral pain and subzonal pain, with scores of 0, 2, 4 and 6 according to the severity. Secondary symptoms include menstrual abdominal pain, fear of cold , loss of appetite, menstrual color, stool, urination, tongue and pulse, etc., tongue and pulse records do not score, other items are given 0, 1, 2, 3 points according to the situation. The higher the total score, the more severe the symptoms.
Local physical sign rating scale | The baseline period, the treatment two menstrual cycle (about 8 weeks) and the follow-up period (about 12 weeks) .
  Local physical sign rating scale included limitation of uterine activity and tenderness, thickening of bilateral appendages and mass, tenderness of bilateral appendages and thickening of uterine-sacral ligament. The score was 0-6. The higher the total score, the more severe the symptoms.
Pelvic masses and fluid accumulation | The baseline period, the treatment two menstrual cycle (about 8 weeks) and the follow-up period (about 12 weeks) .
  Pelvic mass was evaluated according to pelvic ultrasound. The original mass disappeared as disappeared; the original mass volume shrank by more than 2/3 compared with that before treatment as significantly reduced; the original mass volume shrank by 1/3-2/3 compared with that before treatment as reduced; the original mass remained unchanged or increased as unchanged or increased. Pelvic fluid was evaluated according to pelvic ultrasound. The original fluid disappeared as disappeared; the original fluid area reduced by more than 2/3 compared with that before treatment as significantly reduced; the original fluid area reduced by 1/3-2/3 compared with that before treatment as reduced; the original fluid remained unchanged or increased as unchanged or increased.
EuroQol Five Dimensions Questionnaire | The baseline period, the treatment two menstrual cycle (about 8 weeks) and the follow-up period (about 12 weeks) .
  The EQ-5D mainly consists of two parts: the EQ-5D Descriptive System and the EQ-5D Visual Analog Scale . In the description section, the EQ-5D will describe the health status in five dimensions: Mobility, Self care, UsualActivities, Pain/Discomfort, and Anxiety/Depression. The questionnaire requires respondents to choose the most suitable option for themselves in each dimension based on their health status. In the evaluation section, respondents used the Visual Analog Scale (EQ-VAS) to assess their overall health status. EQ-VAS records the self rated health status of respondents on a vertical scale. The scale of the ruler is 0-100, where 0 represents "the worst health state you imagine" and 100 represents "the best health state you imagine". The self-assessment information of the respondents can be used as a quantitative indicator of health outcomes.
Recurrence of abdominal pain during 1-month menstrual cycle was followed up. | the treatment two menstrual cycle (about 8 weeks) and the follow-up period (about 12 weeks) .
  Within 1 menstrual cycle after treatment, patients with the main symptom "pain or tingling of lower abdomen" (VAS score was "0") were followed up, and the end point of follow-up was the recurrence point of the main symptoms. If there was no recurrence in one menstrual cycle after the end of treatment, it was the end point of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Master, Principal Investigator — Beijing Hospital of Integrated Traditional Chinese and Western Medicine
Locations (1):
- Beijing Hospital of Integrated Traditional Chinese and Western Medicine, Beijing, China